CLINICAL TRIAL: NCT00579579
Title: Functional Outcomes and Quality of Life in Patients Undergoing Surgery for Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 06-151
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Rectal Cancer
Keywords: Bowel function; Bladder function; Sexual function; Quality of life
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients Undergoing Surgery for Rectal Cancer
  Interventions: Behavioral: Questionaires

INTERVENTIONS:
Behavioral: Questionaires — Prior to surgery, patients will be asked to complete baseline surveys. In addition, a random subsample of approximately 30 patients will be asked to participate in a short qualitative interview to explore expectations regarding bowel function and quality of life following surgery. Follow-up surveys will be completed at 6, 12 and 24 months after bowel continuity has been restored (defined by their last surgical procedure). Patients with a permanent stoma will receive the Stoma-specific QOL questions in place of the MSKCC Bowel Function Instrument at 6 and 12 months after initial surgery.

SUMMARY:
The purpose of this study is to find out what happens to patients after they have surgery for rectal cancer. After being treated for rectal cancer, patients tell us that their bowel, bladder and sexual function have changed. We are trying to understand how these changes affect your quality of life. The research that we have now does not explain these changes or problems very well. The patients will be asked questions about bowel function, bladder function, sexual function, and quality of life so we can understand these changes better. This will help us take better care of our patients in the future, before and after their treatment for rectal cancer.

DETAILED DESCRIPTION:
Rectal cancer is the second most common cancer in North America. Therapy has rapidly improved over the last 20 years, and the surgical technique of total mesorectal excision, as well as advances in radiation and chemotherapy, have resulted in improved survival and decreased local recurrence. As a result, survivorship issues become increasingly important for patients with rectal cancer.

Patients uniformly demonstrate a strong desire to avoid a permanent stoma and show strong preferences for sphincter preserving surgery (SPS). With the introduction of the circular stapler, SPS is technically possible in a higher proportion of patients. Additionally, even tumors at the anorectal ring are considered amenable to SPS in select patients with ultra-low rectal cancers.

At present, long-term outcomes after rectal cancer surgery are poorly understood. Bowel, bladder and sexual function appear to be negatively affected by multi-modality therapy. However, function has been poorly studied, and it is difficult to translate the data into clinically meaningful information for patients. Clinically, bowel, bladder and sexual dysfunction seem to affect quality of life (QOL), although this has never been well studied. It is important to quantify the extent of impairment so that it can be used to educate patients preoperatively. However, translating these data to clinicians and patients remains challenging, and efforts to convey the data in a meaningful manner preoperatively constitute an important element in managing patient expectations. By understanding patients' baseline needs, expectations and satisfaction at the time of the preoperative consent, we can begin to develop novel preoperative strategies for educating patients about postoperative function and quality of life in a meaningful manner, so that they may better adapt after surgery. We ultimately plan to use data from this study to develop and subsequently evaluate the role of an educational tool outlining functional outcomes after rectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III rectal adenocarcinoma based on preoperative testing
* Surgery (Sphincter preserving - transanal (TAE),transanal endoscopic microsurgery (TEM), low anterior resection (LAR), coloanal resection (CAA), OR Permanent stoma - abdominal perineal resection (APR)) planned at MSKCC
* Age > or = to 18
* Speak English

Exclusion Criteria:

* Stage IV disease at time of pre-operative consult
* History of other malignancies (besides squamous cell or basal cell cancer of skin) less than five years ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are being asked to take part in this study because they have rectal cancer and are planning on having surgery done at MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2006-11-28 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
To prospectively evaluate bowel, sexual and bladder function in patients who undergo resection for stage I-III rectal cancer. | Two sets of surveys before surgery. After surgery, the participant will be asked to fill out some or all of a series of surveys at 6, 12, and 24 months.

SECONDARY OUTCOMES:
To assess the impact of bowel, bladder and sexual function on quality of life over time in patients undergoing resection for stage I-III rectal cancer and to compare QOL in patients with and without a stoma. | Two sets of surveys before surgery. After surgery, the participant will be asked to fill out some or all of a series of surveys at 6, 12, and 24 months.
To evaluate the expectations, informational needs and satisfaction with the surgical consent process in patients undergoing resection for stage I-III rectal cancer. | Two sets of surveys before surgery. After surgery, the participant will be asked to fill out some or all of a series of surveys at 6, 12, and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Garcia-Aguilar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org